CLINICAL TRIAL: NCT02965807
Title: Effect of Bronchial Thermoplasty on Moderate Bronchial Asthma in China
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, ShiYue Li, director, Guangzhou Institute of Respiratory Disease
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-17
Record Dates: First submitted 2016-11-09; First posted 2016-11-17 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Moderate Asthma
Keywords: Bronchial Thermoplasty; moderate asthma; China
MeSH Terms: interventions — Bronchial Thermoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bronchial Thermoplasty (Experimental): Moderate bronchial asthma patients under the Bronchial Thermoplasty.
  Interventions: Device: Bronchial Thermoplasty

INTERVENTIONS:
Device: Bronchial Thermoplasty — patients will be under Bronchial Thermoplasty approximately every three weeks.And totally having three surgerys will be considered as completed.

SUMMARY:
This study aims to investigate the efficacy and safety of Bronchial Thermoplasty on moderate bronchial asthma in China, by observing the improvement of quality of life, the decrease of acute attack and emergence, as well as the incidence of related complications.

DETAILED DESCRIPTION:
This is a multi-center, open-label and single arm study. At least 50 patients with moderate asthma receive Bronchial Thermoplasty for three times. Asthma Quality of Life Questionnaire (AQLQ), Asthma Control Questionnaire (ACQ), Frequency of mild asthma acute attack, PEF, FEV1, Emergency and Hospitalization are compared between before and after BT treatment.

The unified peak flow test meter will be provided to all subjects enrolled in this study. They will get a follow-up diary book before leaving hospital. In order to ensure the efficiency, all enrolled asthma patients are trained and tested by doctors and nurses from in-patient or out-patient department when they follow up, including how to use the PEF meter, how to read and record the data. As for the dosage of medication, all the medication uses are followed the doctor's advice, once the rescue medications were used, the times and dosages are mandatory to be recorded in the diary book by the patients themselves.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18y and 65y.
2. no improvement after ICS and LABA treatment in patients with moderate asthma
3. have not received BT before
4. stable more than 6 weeks before enrolled in this study
5. no implantable electrical device (e.g. cardiac pacemaker)
6. no permanent anticoagulant is being used

Exclusion Criteria:

1. Smoking and have obvious emphysema
2. Chest CT showed lower lobe bronchial stenosis or distal complete atelectasis
3. FEV1 < 65% predicted value after using bronchodilator
4. airway infection(within 6 weeks)
5. any circumstances as the following within the past 1 year: lower respiratory tract infection (LRTI) for 4 times or above; hospitalization due to respiratory diseases for more than 3 times; increase the dosage of oral corticosteroids due to asthma exacerbation for more than 4 times
6. received endotracheal intubation or ICU admission due to asthma attack within the past 2 years
7. concomitant allergic bronchopulmonary aspergillosis
8. Implantable electronic devices (such as cardiac pacemaker)/NYHA class IV and/or acute myocardial infarction within the past 3 months
9. coagulation disorders,cannot stop taking anticoagulant、antiplatelet drugs or nonsteroidal anti-inflammatory drugs
10. increasing the risk of adverse reactions during bronchoscopy or anesthesia as the followings: pregnancy, insulin-dependent diabetes, epilepsy, or the other severe complications, such as uncontrolled coronary heart disease, acute or chronic renal failure or uncontrolled hypertension
11. others:vocal cord dysfunction、chronic nasosinusitis、airway obstruction or uncontrolled obstructive sleep apnea syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
change from baseline2 AQLQ score after Bronchial Thermoplasty | baseline2、6 weeks after the third surgery、3、6、9 、12 months after the third surgery and stoping laba for 2 weeks

SECONDARY OUTCOMES:
decline from baseline 2 in the ACQ score for 0.5 or more | baseline2、6 weeks after the third surgery、3、6、9 、12 months after the third surgery and stoping laba for 2 weeks
Frequency of mild asthma acute execration after Bronchial Thermoplasty | baseline2、6 weeks after the third surgery、3、6、9 、12 months after the third surgery and stoping laba for 2 weeks
  A mild exacerbation is defined as 2 consecutive days when at least one of the following occurs:1. Morning peak expiratory flow falls at least 20% below the average morning peak flow recorded at the baseline (the first 2 weeks during the 4-week baseline period).
  2. More than 3 more puffs of rescue short acting bronchodilator are required than the average usage at the baseline(the first 2 weeks during the 4-week baseline period).
  3. Awakening at night with asthma symptoms.
change from baseline2 peak flow after Bronchial Thermoplasty | baseline2、6 weeks after the third surgery、3、6、9 、12 months after the third surgery and stoping laba for 2 weeks
change from baseline2 FEV1 after Bronchial Thermoplasty | baseline2、6 weeks after the third surgery、3、6、9 、12 months after the third surgery and stoping laba for 2 weeks
change from baseline2 FEV1/FVC after Bronchial Thermoplasty | baseline2、6 weeks after the third surgery、3、6、9 、12 months after the third surgery and stoping laba for 2 weeks
change from baseline2 FEV1 predicted after Bronchial Thermoplasty | baseline2、6 weeks after the third surgery、3、6、9 、12 months after the third surgery and stoping laba for 2 weeks
the percentage of Emergency | baseline2、6 weeks after the third surgery、3、6、9 、12 months after the third surgery and stoping laba for 2 weeks
Hospitalization and Asymptomatic days | baseline2、6 weeks after the third surgery、3、6、9 、12 months after the third surgery and stoping laba for 2 weeks
the incidence of severe respiratory adverse events | baseline2、6 weeks after the third surgery、3、6、9 、12 months after the third surgery and stoping laba for 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: shiyue li, director, Principal Investigator — Guangzhou Institute of Respiratory Disease
Locations (1):
- Guangzhou Institute of Respiratory Disease, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Solway J, Irvin CG. Airway smooth muscle as a target for asthma therapy. N Engl J Med. 2007 Mar 29;356(13):1367-9. doi: 10.1056/NEJMe078005. No abstract available. PMID 17392308
- [Background] Danek CJ, Lombard CM, Dungworth DL, Cox PG, Miller JD, Biggs MJ, Keast TM, Loomas BE, Wizeman WJ, Hogg JC, Leff AR. Reduction in airway hyperresponsiveness to methacholine by the application of RF energy in dogs. J Appl Physiol (1985). 2004 Nov;97(5):1946-53. doi: 10.1152/japplphysiol.01282.2003. Epub 2004 Jul 16. PMID 15258133
- [Background] Lai CK, De Guia TS, Kim YY, Kuo SH, Mukhopadhyay A, Soriano JB, Trung PL, Zhong NS, Zainudin N, Zainudin BM; Asthma Insights and Reality in Asia-Pacific Steering Committee. Asthma control in the Asia-Pacific region: the Asthma Insights and Reality in Asia-Pacific Study. J Allergy Clin Immunol. 2003 Feb;111(2):263-8. doi: 10.1067/mai.2003.30. PMID 12589343
- [Result] Miller JD, Cox G, Vincic L, Lombard CM, Loomas BE, Danek CJ. A prospective feasibility study of bronchial thermoplasty in the human airway. Chest. 2005 Jun;127(6):1999-2006. doi: 10.1378/chest.127.6.1999. PMID 15947312
- [Result] Cox G, Thomson NC, Rubin AS, Niven RM, Corris PA, Siersted HC, Olivenstein R, Pavord ID, McCormack D, Chaudhuri R, Miller JD, Laviolette M; AIR Trial Study Group. Asthma control during the year after bronchial thermoplasty. N Engl J Med. 2007 Mar 29;356(13):1327-37. doi: 10.1056/NEJMoa064707. PMID 17392302
- [Result] Pavord ID, Cox G, Thomson NC, Rubin AS, Corris PA, Niven RM, Chung KF, Laviolette M; RISA Trial Study Group. Safety and efficacy of bronchial thermoplasty in symptomatic, severe asthma. Am J Respir Crit Care Med. 2007 Dec 15;176(12):1185-91. doi: 10.1164/rccm.200704-571OC. Epub 2007 Sep 27. PMID 17901415
- [Result] Castro M, Rubin A, Laviolette M, Hanania NA, Armstrong B, Cox G; AIR2 Trial Study Group. Persistence of effectiveness of bronchial thermoplasty in patients with severe asthma. Ann Allergy Asthma Immunol. 2011 Jul;107(1):65-70. doi: 10.1016/j.anai.2011.03.005. Epub 2011 Apr 14. PMID 21704887
- [Result] Cox G, Miller JD, McWilliams A, Fitzgerald JM, Lam S. Bronchial thermoplasty for asthma. Am J Respir Crit Care Med. 2006 May 1;173(9):965-9. doi: 10.1164/rccm.200507-1162OC. Epub 2006 Feb 2. PMID 16456145